CLINICAL TRIAL: NCT00041353
Title: Breast Cancer Biomarkers Based on Fine Needle Aspirates
Brief Title: Comparison of Biomarkers Based on Fine-Needle Aspiration in Women at Increased or Normal Risk of Breast Cancer
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was not activated at Fox Chase Cancer Center
Sponsor: Fox Chase Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Screening
Other Study IDs: FCCC-02010; CDR0000069491 (Registry Identifier: PDQ (Physician Data Query)); NCI-G02-2095
Record Dates: First submitted 2002-07-08; First posted 2003-05-26 (Estimated); Last update posted 2013-07-11 (Estimated); Status verified 2013-07

CONDITIONS: Breast Cancer
Keywords: ductal breast carcinoma in situ; lobular breast carcinoma in situ
MeSH Terms: conditions — Breast Neoplasms; Carcinoma, Intraductal, Noninfiltrating; Breast Carcinoma In Situ

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: cytology specimen collection procedure
Procedure: comparison of screening methods
Procedure: study of high risk factors

SUMMARY:
RATIONALE: Examining biomarkers in fine-needle aspiration specimens from women at risk for breast cancer may improve the ability to detect breast cancer cells early and plan effective treatment.

PURPOSE: Screening trial to compare specific biomarkers based on fine-needle aspiration specimens from women at increased or normal risk of breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare specific biomarkers, including cellular morphology (cytology), proliferation index (Ki-67), p53 expression, and LOH in chromosome 9p at locus DS9157, in fine needle aspirate specimens from women at increased vs normal risk of breast cancer.
* Determine whether these specimens are adequate to perform the biomarker assays and whether this technique could be used in the general outpatient setting.
* Determine whether biomarker levels in these patients are concordant or discordant with individual clinical risk of breast cancer.
* Determine whether 1 or more biomarkers can distinguish high-risk from control patients.
* Correlate specific biomarkers and changes in biomarker levels with pathologic diagnosis from the breast biopsy.

OUTLINE: Patients undergo fine needle aspiration of normal appearing breast tissue prior to the beginning of elective surgery. Specimens are analyzed for the presence of specific biomarkers.

PROJECTED ACCRUAL: Approximately 156 patients will be accrued for this study within 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Increased risk of breast cancer as determined by 1 or more first-degree relatives (mother, sister, or daughter) with a history of breast cancer OR a personal history of atypical hyperplasia, lobular carcinoma in situ, or ductal carcinoma in situ of the breast OR
* No increased risk of breast cancer as determined by a lack of the above conditions
* Scheduled to undergo elective breast surgery for removal of a mammographic lesion or palpable breast lump
* No prior bilateral mastectomy or bilateral breast irradiation
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Age:

* 30 and over

Sex:

* Female

Menopausal status:

* Not specified

Performance status:

* Not specified

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* Not specified

Renal:

* Not specified

Other:

* No active invasive malignancy in any site except basal cell or squamous cell skin cancer
* No significant medical or psychiatric problems that would preclude study
* No evidence of excessive use of narcotics or drug dependency

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* Not specified

Endocrine therapy:

* Not specified

Radiotherapy:

* See Disease Characteristics

Surgery:

* See Disease Characteristics

Min Age: 30 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Primary Completion 2002-09 (Actual); Study Completion 2002-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael H. Torosian, MD, Study Chair — Fox Chase Cancer Center